CLINICAL TRIAL: NCT06516848
Title: High-intensity Inspiratory Muscle Training in Patients With Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Assoc.Dr., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Asthma_IMT
Record Dates: First submitted 2024-07-04; First posted 2024-07-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Asthma
Keywords: inspiratory muscle training; exercises
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Inspiratory Muscle Training Group (H-IMT) (Experimental)
  Interventions: Other: High Intensity Inspiratory Muscle Training Group (H-IMT)
- Low Intensity Inspiratory Muscle Training Group (L-IMT) (Experimental)
  Interventions: Other: Low Intensity Inspiratory Muscle Training Group (L-IMT)

INTERVENTIONS:
Other: High Intensity Inspiratory Muscle Training Group (H-IMT) — Respiratory muscle strengthening training will be given with a resistive threshold inspiratory muscle strengthening device. Initially, it will be worked out vigorously at 80% of the maximum inspiratory pressure determined by mouth pressure measurement. The load will be increased weekly.
  Arms: High Intensity Inspiratory Muscle Training Group (H-IMT)
Other: Low Intensity Inspiratory Muscle Training Group (L-IMT) — Respiratory muscle strengthening training will be given with a resistive threshold inspiratory muscle strengthening device. Initially, it will be worked out vigorously at 30% of the maximum inspiratory pressure determined by mouth pressure measurement. The load will be increased weekly.
  Arms: Low Intensity Inspiratory Muscle Training Group (L-IMT)

SUMMARY:
The aim of this study is to examine the effects of high-intensity and low-intensity inspiratory muscle training added to the standard pulmonary rehabilitation exercise program including aerobic and peripheral muscle strengthening training on respiratory muscle function, exercise capacity, dyspnea and health-related quality of life in asthmatic patients. The aim of the study was to examine whether there are intra-group changes and inter-group differences in the groups where low and high intensity inspiratory muscle training was applied. The cases meeting the inclusion criteria will be randomized and divided into two groups, the groups will be named as High Intensity Inspiratory Muscle Training Group (H-IMT) and Low Intensity Inspiratory Muscle Training Group (L-IMT).

DETAILED DESCRIPTION:
Patients diagnosed with asthma by a chest diseases specialist and referred to pulmonary rehabilitation will be included in the study. The cases meeting the inclusion criteria will be randomized and divided into two groups, the groups will be named as High Intensity Inspiratory Muscle Training Group (H-IMT) and Low Intensity Inspiratory Muscle Training Group (L-IMT). Inspiratory muscle training will be carried out in the form of 2 minutes of work and 1 minute break for a total of 21 minutes, starting from 80% of the maximum inspiratory pressure determined by mouth pressure measurement for the H-IMT Group and 30% for the L-IMT Group. An 8-week training will be carried out by increasing the planned load by 5% every two weeks. In addition, breathing exercises, strengthening exercises and walking training on flat ground will be given to both groups in the form of a home program. The training program will be 8 weeks in total, 3 days a week. will be given online exercises, synchronized 2 days a week, and a home program for 1 day, accompanied by a physiotherapist, via videoconference on the smartphone. A total of 24 sessions will be held.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65 years
* Having been diagnosed with severe persistent, non-allergic asthma by a pulmonologist in accordance with the Global Initiative for Asthma (GINA) guideline criteria,
* Patients with type 2 inflammation markers. According to accepted standards; peripheral eosinophils <150/µL and/or negative skin prick test and/or total IgE <30 kU/L
* Bronchodilator response (>12% or 200 mL improvement in FEV1% predicted following inhalation of 400 mg salbutamol)
* Those who were diagnosed at least 6 months ago and are under follow-up and treatment, and/or patients whose asthma is under control

Exclusion Criteria:

* Having recently had a respiratory tract infection recently (within the last month),
* Having a smoking history of more than 10 pack-years or having a history of smoking within 6 months after quitting smoking
* Having received oral corticosteroid treatment in the last 4 weeks,
* Having a Body Mass Index >35,
* Eosinophilic Granulomatosis Polyangiitis (EGPA) and Allergic Bronchopulmonary Aspergillosis (ABPA),
* Vasculitis,
* History of malignancy,
* Pregnancy,
* Previous lung surgery, use of long-term oxygen therapy
* Having accompanying restrictive lung diseases (advanced kyphoscoliosis, ankylosing spondylitis) and neuromuscular diseases (myasthenia gravis, muscular dystrophies, myopathies) that will prevent healthy respiratory function testing and rehabilitation.
* Having conditions such as cognitive dysfunction, mental retardation, dementia that make it difficult to implement the protocol or interpret the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) measurement | Change from baseline respiratory muscle strength at 8 weeks
  Respiratory muscle strength will be assessed via maximal inspiratory pressure (MIP). Tests will be carried out according to American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria.
Six minute walking test | Change from baseline 6 minute walking distance at 8 weeks
  The exercise capacity will be assessed by the 6-minute walking test. The test will be conducted in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines.
Modified Medical Research Council (mMRC) Dyspnea Scale | Change from baseline dyspnea perception at 8 weeks
  The Modified Medical Research Council (mMRC) Dyspnea Scale will be used to evaluate the patients' dyspnea levels. The mMRC will consist of a 0-4 point category scale in which the patient will choose the statement that best describes their dyspnea level among 5 statements that express the feeling of difficulty in breathing experienced in daily life activities. A higher score will indicate greater dyspnea severity.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | Change from baseline FVC at 8 weeks
  Pulmonary function test will be performed using the Pony Fx spirometry device, according to the American Thoracic Society (ATS) guidelines. FVC is the volume of air that can forcibly be blown out after full inspiration.
Forced Expiratory Volume (FEV1) | Change from baseline FEV1 at 8 weeks
  Change in Forced Expiratory Volume (FEV1) will be measured using spirometry as the maximal volume of air (liters) exhaled in the first second of expiration.
Peak Expiratory Flow (PEF) | Change from baseline PEF at 8 weeks]
  Change in Peak Expiratory Flow (PEF) will be measured using spirometry as the maximal speed of expiration (measured in liters/min).
FEV1/FVC | Change from baseline FEV1/FVC at 8 weeks]
  Spirometry will be used to measure the values of FEV1/FVC three times. The highest result will be recorded.
Asthma Control Test (ACQ) | Change from baseline ACQ score at 8 weeks
  The ACQ will be a test that allows subjective evaluation of the last 4 weeks of disease control in asthma patients. The ACQ will consist of 5 items that the patient can complete themselves. Each item will be scored between 1 and 5. An ACQ score of 25 will indicate "controlled" asthma, a score between 20 and 24 will indicate "partially controlled" asthma, and a score <20 will indicate "uncontrolled" asthma.
Peripheral muscle strength | Change from baseline peripheral muscle strength at 8 weeks
  Peripheral muscle strength will be assessed by a hand-held dynamometer.
Asthma Quality of Life Scale (AQLQ) | Change from baseline AQLQ score at 8 weeks]
  This survey will consist of 32 questions in four disease-specific health areas. The AQLQ will include 12 questions about symptoms, 11 questions about limitations in activities, 5 questions about emotional state, and 4 questions about environmental stimuli. Patients will be asked to respond to each item on a 7-point scale (1: Severe impairment, 7: No impairment) considering their quality of life in the last two weeks. The total score average and average scores for sub-dimensions will be calculated. The average of the obtained values will be evaluated between 1 and 7.
St. George Respiratory Questionnaire (SGRQ) | Change from baseline SGRQ score at 8 weeks
  This will be a self-administered questionnaire that can be completed by the patient to determine disease-specific quality of life. The test will consist of 50 items divided into 3 parts measuring the symptoms of the disease, activity limitation, and social/emotional impact. The activity component will relate to physical activities that may cause or are limited by shortness of breath. The impact component will include factors such as work, occupation, medications taken to keep one's health under control, side effects of medications, difficulty in continuing daily life activities, and panic. The three parts of the test will be scored separately and the total score will be calculated. St. George Respiratory Questionnaire scores will range from 0 (no impairment in quality of life) to 100 (poor quality of life). In the SGRQ questionnaire, a change of four units due to treatment will be considered significant.
International Physical Activity Questionnaire- short form | Change from baseline physical activity level at 8 weeks
  Physical activity level will be assessed by the International Physical Activity Questionnaire - Short Form. This will include seven questions on the frequency and duration of time spent in physical activity in the past 7 days to calculate a score for each domain (walking, moderate-intensity activities, and vigorous-intensity activities) and an overall grand total expressed in MET-minutes/week. MET values and formula for computation of MET-minutes: Walking MET-minutes/week = 3.3 * walking minutes * walking days; Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days; Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days. A combined total physical activity MET-min/week will be computed as the sum of Walking + Moderate + Vigorous MET-min/week scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehli̇van, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kocak C, Pehlivan E, Baslilar S. High- vs. low-intensity inspiratory muscle training in asthma: effects on respiratory muscles, exercise performance, dyspnea, and health-related quality of life. J Asthma. 2025 Oct;62(10):1776-1788. doi: 10.1080/02770903.2025.2519103. Epub 2025 Jun 20. PMID 40524414